CLINICAL TRIAL: NCT00506246
Title: A Multi-Center, Randomized, Double-Blind, Positive Controlled Study to Evaluate the Efficacy and Safety of Propofol(Propofol®-Lipuro) in Total Intravenous Anaesthesia
Brief Title: Efficacy and Safety Study of Two Propofol Formulations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Collaborators: B. Braun Medical International Trading Company Ltd. (Industry); Tigermed Consulting Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006L00667
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2008-02

CONDITIONS: General Anaesthesia; Induction of Anaesthesia
Keywords: anaesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Propofol MCT/LCT
  Interventions: Drug: Propofol
- 2 (Active Comparator): Propofol LCT
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — * intravenous (total intravenous anaesthesia)
  * induction and maintenance
  Other Names: Propofol Lipuro 1%; Diprivan 1%

SUMMARY:
The purpose of the study to compare Propofol-MCT/LCT with LCT in terms of their efficacy and safety during total intravenous anaesthesia

DETAILED DESCRIPTION:
Propofol (chemical substance 2, 6-Diisopropylphenol) is a short-acting intravenous general anaesthetic which is used for induction and maintenance of a general anaesthesia, for long-term sedation of ventilated intensive care patients or for short-term sedation in diagnostic and surgical procedures. As an active substance propofol produces good and readily controlled anaesthesia with smooth and problem-free recovery both in adult patients and in children over 1 month of age. One potential advantage of this formulation is that the MCT/LCT-emulsion reduces pain on injection, a frequently reported adverse reaction with LCT-emulsions of propofol.

ELIGIBILITY:
Inclusion Criteria:

* Female and male adult patients, and at least 18 and maximal 65 years of age;
* ASA-classification I to II;
* Undergoing an elective surgery, the anaesthesia is expected to last at least 1 hour and no more than 3 hours;
* Will be under total intravenous anaesthesia;
* Willing to give their signed informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
time to loss of eyelash reflex | induction of anaesthesia
doses required for induction of anaesthesia until loss of eyelash reflex | induction of anaesthesia

SECONDARY OUTCOMES:
patient data/history | during anaesthesia
pre- and concomitant medication | during anaesthesia
anaesthesia relating data | during anaesthesia
recovery data | during anaesthesia
drug safety data (e.g. haemodynamics and clinical outcome) | during anaesthesia
adverse events | during anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Zhanggang Xue, Prof, Principal Investigator — Shanghai Zhongshan Hospital
Locations (3):
- China (3):
  - Pekin Union Medical College Hospital, Beijing
  - Renji Hospital Affiliated to Shanghai Jiaotong University, Shanghai
  - Zhongshan Hospital affiliated to Fudan University, Shanghai